CLINICAL TRIAL: NCT05803616
Title: Liquid Biopsy-based Genomic Assay to Enable Non-invasive Precision Diagnostics and Monitoring for Immune-mediated Lymphoproliferative Disorders (ILD)
Brief Title: Liquid Biopsy to Enable Diagnostics and Monitoring for Immune-mediated Lymphoproliferative Disorders
Acronym: LIMPID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Noémie Lang, DR, University Hospital, Geneva
Other Study IDs: 2021-01016
Record Dates: First submitted 2023-03-09; First posted 2023-04-07 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Lymphoproliferative Disorders; Lymphoproliferative Disorder Following Transplantation
Keywords: Immune-related Lymphoproliferative Disorders
MeSH Terms: conditions — Lymphoproliferative Disorders | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood 20 ml at each time point defined as per protocol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ILD group: All patients newly diagnosed or relapsing from an ILD could be enrolled in this observational study
  Interventions: Diagnostic Test: Liquid biopsy

INTERVENTIONS:
Diagnostic Test: Liquid biopsy — ctDNA measured in the plasma and analyse by next generation sequencing (NGS) for minimal residual disease (MRD)

SUMMARY:
Immune-mediated lymphoproliferative disorders (ILD), as per World Health Organization (WHO HAEM 5) classification, are rare conditions associated with a poor outcome. Current management of ILD is focusing on prevention (e.g.) early detection of ILD with preemptive Epstein Barr virus (EBV) Deoxyribonucleic acid (DNA) levels monitoring, however, this approach is useless for the early detection of EBV-negative ILD. Therapeutic management consists of a reduction in immunosuppressive therapy (RIS), allowing mostly partial and transient responses. Rituximab, an anti-CD20 (cluster differentiation 20) antibody, provides roughly 20-25% of complete and durable responses, thus the majority of ILD patients will require immunochemotherapy, burden with significant toxicity in this challenging population. Implementation of liquid biopsy, also called circulating tumor DNA (ctDNA) in plasma or serum is an area of investigation that is becoming increasingly relevant for clinical practice, allowing for non-invasive monitoring of disease status.

Early detection and monitoring of ILD using ctDNA may allow for preemptive therapy, improved risk-stratification and ultimately, lead to outcome improvement. This multicenter Swiss project will allow a better understanding of ILD mutational landscape and pathogenesis, which could lead to the development of new screening and monitoring approaches for patients suffering from ILD.

DETAILED DESCRIPTION:
In this observational prospective study, the investigators will collect clinical data from subjects' charts through a dedicated multicenter electronic case report form (eCRF).

Whenever available, PET-CT will be transferred through a Web-based Imaging and Diagnosis Exchange Network (WIDEN) to perform a blinded independent review of staging and response.

Biological samples included 20 ml of blood collected at each of the following planned clinical points in time: i) at ILD diagnosis, ii) after first cycle of therapy, iii) at interim response assessment, iv) at the end-of-treatment, v) at 3 months follow-up, vi) at 12 months follow-up, vii) at disease progression, if applicable. Additional samples could be collected if clinically relevant.

Additionally, the investigators will request formalin-fixed and paraffin-embedded tissue (FFPET) or fresh-frozen (FF) tissue slices/blocks at ILD diagnosis from Pathology Departments of participating Centers for retrospective ILD subjects.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a diagnosis of ILD defined by the World Health Organization (WHO HAEM 5)(e.g. post-transplant setting, X-link, concomitant auto-immune disorders)

Exclusion Criteria:

* Lymphoproliferative disorders non immune-mediated
* Lymphoproliferative disorders occurring in the context of a concomitant human immunodeficiency virus (HIV) infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients newly diagnosed or relapsing from an ILD as per World Health Organization (WHO HAEM 5) classification
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive value of ctDNA to monitor response in ILD (MRD) using NGS | 2 years
  Molecular response (minimal residual disease, MRD) during therapy in ILD diagnosed patients will be monitored using regular liquid biopsy (ctDNA) and assessing the presence or not of genomic aberrations present at baseline if any.

SECONDARY OUTCOMES:
Characterisation of ILD tumour microenvironment and genetic / epigenetic landscape | 2 years
  Tumour microenvironment and genetic / epigenetic landscape will be explored using various techniques such as NGS, multiplex immunohistochemistry, digital droplet Polymerase Chain Reaction (ddPCR) and methyloma assays.

CONTACTS AND LOCATIONS:
Overall Officials: Noemie Lang, MD, Principal Investigator — Geneva Univresity Hospital
Locations (6):
- Switzerland (6):
  - Basel University Hospital, Basel
  - Oncology Institute of Southern Switzerland, Bellinzona
  - Inselspital, Bern
  - Hôpitaux Universitaires de Genève (HUG), Geneva
  - Kantonsspital, Sankt Gallen
  - University Hospital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
All anonymised IPD that underlie results in a publication will be shared upon request with other researchers.
  Types of supporting information that will be shared, in addition to the individual participant data set and data dictionaries will include the study protocol, informed consent form and clinical study report
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available one month after study results publication with no limit of time.
Access Criteria: All data supporting the findings of the current study will be made available from the corresponding author upon reasonable scientific request